CLINICAL TRIAL: NCT03640429
Title: Accuracy and Trending of Non-invasive Oscillometric Blood Pressure Monitoring at the Wrist in Obese Patients
Brief Title: Accuracy of Non-invasive Blood Pressure Monitoring at the Wrist in Obese Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Other Study IDs: N-72-2018
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Blood Pressure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: non-invasive blood pressure monitor — non-invasive oscillometric blood pressure monitor will be applied at the arm, forearm, and at the wrist.
Device: invasive blood pressure monitor — invasive blood pressure monitor will be connected to a cannula inserted at the radial artery.

SUMMARY:
Arterial blood pressure (ABP) monitoring is a corner stone in perioperative management. However, proper control of SBP requires accurate measurement of ABP.

The aim of this work is to validate the wrist OBP monitor in obese patients and compare it to upper arm location (in accuracy, convenience, and trending) using invasive blood pressure monitor as a reference standard.

DETAILED DESCRIPTION:
Arterial blood pressure (ABP) monitoring is a corner stone in perioperative management. Recently, tight intraoperative individualized control of systolic blood pressure (SBP) (within 10% of baseline reading) was reported to reduce the risk of postoperative organ dysfunction in high risk patients undergoing abdominal procedures. However, proper control of SBP requires accurate measurement of ABP.

The gold standard for ABP measurement is through a catheter placed in an artery. Being an invasive, measurement of BP through an arterial catheter is restricted to patients with rapid major fluid shifts. Many indirect methods are used for measurement of ABP. Oscillometric blood pressure (OBP) monitoring is considered the standard non-invasive monitor for use in most clinical situations. In OBP monitor, a pressure transducer located in the cuff senses the series of small oscillations heart-beat induced pulse volume changes. These oscillations are detected during deflation of the cuff pressure from above the SBP to diastolic blood pressure (DBP).

The upper arm is the standard location of application of the blood pressure cuff as it is aligned with the heart level regardless the patient position. In obese patients, OBP monitoring is considered superior to auscultatory method which is limited by faint auscultatory sounds. However, application of blood pressure cuff at the upper arm in this population is frequently limited by large arm circumference and asymmetrical arm contour. Thus, locating the cuff at the wrist might be a more feasible alternative for the upper arm. OBP monitoring at the wrist was previously compared to auscultatory measurement of ABP in non-surgical patients. A recent study investigated the accuracy of OBP at the upper forearm in obese patients. No data to the best of our knowledge validated OBP monitoring at the lower forearm in obese patients using invasive blood pressure monitor as a reference standard.

The aim of this work is to validate the wrist OBP monitor in obese patients and compare it to upper arm location (in accuracy, convenience, and trending) using invasive blood pressure monitor as a reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged above 18 years)
* obese (with body mass index above 30 Kg/squared meter)

Exclusion Criteria:

* Peripheral vascular diseases
* Upper limb operations
* Upper limb scars
* Upper limb deep venous thrombosis
* Arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, obese, patients scheduled to surgery under general anesthesia will be included in the study. Arterial catheter will be inserted and used as a reference for evaluation of non-invasive blood pressure monitor at different sites.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 hours
  Systolic blood pressure measured in mmHg

SECONDARY OUTCOMES:
Diastolic blood pressure | 3 hours
  Systolic blood pressure measured in mmHg
mean blood pressure | 3 hours
  Mean blood pressure measured in mmHg
Heart rate | 3 hours
  The number of heart beats per minute
Body mass index | 5 minutes
  The ratio between the body weight and height of the patient measured by Kg per squared meter
Arm circumference | 5 minutes
  The circumference of the arm measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, Professor, Principal Investigator — Assistant professor of anesthesia
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No